CLINICAL TRIAL: NCT01513096
Title: Efficacy of Prokinetics With Split Dose of PEG in Morning Colonoscopic Bowel Preparation: A Randomized, Controlled Trial
Brief Title: Efficacy of Prokinetics With Split Dose of PEG in Morning Colonoscopic Bowel Preparation
Acronym: PSPEG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, MD, Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: GI-201201
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-01

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: colonoscopy; bowel preparation; PEG; Prokinetics
MeSH Terms: interventions — itopride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Split-dose PEG (No Intervention): Bowel preparation using split dose PEG without prokinetics
- Split dose PEG with prokinetics (Active Comparator): Bowel preparation using split-dose PEG with prokinetics
  Interventions: Drug: itopride

INTERVENTIONS:
Drug: itopride — itopride, 10mg, twice per day, for 1 day
  Arms: Split dose PEG with prokinetics

SUMMARY:
In bowel preparation using split dose PEG, various adjuncts to colonic cleansing were proposed to improve colonic preparation cleansing. Prokinetics, as an adjunct, was included in a few studies. The investigators study was to show that sufficient dosage of prokinetics added to split dose of PEG improves the state of bowel preparation.

DETAILED DESCRIPTION:
This was a randomized, prospective, endoscopist-blinded clinical trial in which the efficacy of prokinetics coadministrated with split dose PEG on the bowel cleansing was inspected.

Endoscopists, who were blinded to the study group of the patient, immediately completed the Ottawa scale and the fluidity scale after procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient who are scheduled for colonoscopy

Exclusion Criteria:

* pregnancy,
* breast feeding,
* known or suspected bowel obstruction, and
* known allergy to PEG or Itopride ,
* presence of severe illness(renal failure, congestive heart failure, liver failure,), and
* refusal of consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
bowel cleaning quality according to Ottawa scale scores | 3 months

SECONDARY OUTCOMES:
procedure time and polyp detection rate | 3 months
  cecal intubation time, polyp detection rate, degree of patient discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Haeundae Paik Hospital, Inje University School of Medicine, Busan, South Korea